CLINICAL TRIAL: NCT04304924
Title: Motivating to Exercise and Diet, and Educating to Healthy Behaviors After Breast Cancer
Acronym: MEDEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-A02374-53; 2019/2986 (Other: CSET number)
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Overweight or Obese Breast Cancer Patients
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial that compares two weight loss programs (control health education program vs. personalized telephone-based health education program) for overweight patients with early breast cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised telephone-based health education (Experimental): The personalized telephone based intervention:
  1. Provide Behavioral support to facilitate lifestyle change by a weight loss coach located at a centralized call center. Participants will be paired with an individual coach who will work with the participant through all phases of the 1-year weight loss program. The behavior change program will be based on Social Cognitive Theory, which hypothesizes that the interactions between environmental, personal and behavioral elements determine behavioral change (Bandura 1989);
  2. Utilize a toolbox approach that will allow for tailoring the intervention to the individual participant. Examples of possible Toolbox solutions include: alternative dietary approaches, instructions for strength-training exercises.
  Interventions: Other: The personalized telephone based intervention
- Standard health educational program (No Intervention)

INTERVENTIONS:
Other: The personalized telephone based intervention — The personalized telephone based intervention:
  1. Provide Behavioral support to facilitate lifestyle change by a weight loss coach located at a centralized call center. Participants will be paired with an individual coach who will work with the participant through all phases of the 1-year weight loss program. The behavior change program will be based on Social Cognitive Theory, which hypothesizes that the interactions between environmental, personal and behavioral elements determine behavioral change (Bandura 1989);
  2. Utilize a toolbox approach that will allow for tailoring the intervention to the individual participant. Examples of possible Toolbox solutions include: alternative dietary approaches, instructions for strength-training exercises.
  Arms: Personalised telephone-based health education

SUMMARY:
The primary objective of MEDEA is to compare the effect of a personalised telephone-based health education weight loss program based on motivational coaching, exercise and diet versus a standard health educational program control on fatigue of overweight or obese BC patients (as measured by the EORTC QLQ C30 (Aaronson et al. 1993; Sprangers et al. 1996))

ELIGIBILITY:
Inclusion Criteria:

This study will be focused on an overweight/obese (BMI ≥25 kg/m2) population of patients with early BC. Particularly, patients will be eligible if they have:

* Documentation of Disease:

  1. Subjects must have histologically confirmed invasive BC and registration must occur within 12 months after the end of active treatment,
  2. Bilateral breast carcinoma is allowed,
  3. Patients must have Stage I toIII BC and no evidence of distant metastatic or locally recurrent disease,
  4. No history of invasive BC in 5 years prior to study registration other than the current diagnosis (prior Ductal Carcinoma in situ (DCIS) at any time does not make a patient ineligible).
* Documentation of overweight/obesity: Subjects must have a BMI ≥25 kg/m2 objectively assessed at the time of eligibility evaluation or reported in the medical records within 56 days prior to study registration. The most recent BMI obtained must be used for eligibility. If most recent BMI is <25 then the patient is not eligible to enroll.
* Prior Treatment :

  1. All adjuvant or neoadjuvant CT, radiation, and surgery completed at least 21 days prior to registration to a maximum of 365 days after the end of treatment,
  2. Patients may have breast reconstruction during protocol participation, but definitive BC surgery must be completed at least 21 days prior to registration,
  3. Biologic therapy, hormonal therapy, and bisphosphonates are acceptable.
* Other:

  1. Age ≥ 18 years,
  2. ECOG Performance Status 0 or 1,
  3. Self-reported ability to walk at least 400 metres (at any pace),
  4. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol,
  5. Patients must be affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product that has Fatigue as a known frequent adverse effects during the last 3 months and while on study treatment,
2. Participating in another weight loss, physical activity or dietary intervention clinical trial. Participants in both arms are also allowed to pursue weight loss and physical activity programs on their own, as long as these programs are not provided as part of a clinical trial,
3. Comorbid conditions, such as other malignancy, diabetes, inflammatory bowel disease, history of severe cardiovascular, respiratory or musculoskeletal disease that would preclude adherence to the study diet or physical activity program or significantly affect the physical status, or the ability to give an informed consent,
4. Secondary overweight or obesity documented or suspected,
5. Chronic consumption of corticosteroids,
6. Self reported pregnancy or intent to become pregnant in the year after enrollement,
7. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Fatigue | up to 12 months
  will be assessed using the EORTC QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Meglio A, Martin E, Crane TE, Charles C, Barbier A, Raynard B, Mangin A, Tredan O, Bouleuc C, Cottu PH, Vanlemmens L, Segura-Djezzar C, Lesur A, Pistilli B, Joly F, Ginsbourger T, Coquet B, Pauporte I, Jacob G, Sirven A, Bonastre J, Ligibel JA, Michiels S, Vaz-Luis I. A phase III randomized trial of weight loss to reduce cancer-related fatigue among overweight and obese breast cancer patients: MEDEA Study design. Trials. 2022 Mar 4;23(1):193. doi: 10.1186/s13063-022-06090-6. PMID 35246219